CLINICAL TRIAL: NCT01180179
Title: Prevention of Recurrent Idiopathic Gastroduodenal Ulcer Bleeding: a Double-blind Randomized Trial
Brief Title: PPI vs H2RA in Patients With Helicobacter Pylori-Negative Idiopathic Bleeding Ulcers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Francis KL Chan, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NNH_RCT
Record Dates: First submitted 2010-08-03; First posted 2010-08-12 (Estimated); Last update posted 2019-08-01 (Actual); Status verified 2019-07

CONDITIONS: Peptic Ulcer
Keywords: H. pylori-negative idiopathic peptic ulcers; Recurrent ulcer bleeding
MeSH Terms: conditions — Peptic Ulcer | interventions — Lansoprazole; Famotidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lansoprazole 30mg once daily (Active Comparator): Lansoprazole 30mg once daily
  Interventions: Drug: Lansoprazole
- Famotidine 40mg once daily (Active Comparator): Famotidine 40mg once daily
  Interventions: Drug: Famotidine

INTERVENTIONS:
Drug: Lansoprazole — 30mg once daily
  Arms: Lansoprazole 30mg once daily
Drug: Famotidine — 40mg once daily
  Arms: Famotidine 40mg once daily

SUMMARY:
The aim of this study is to compare the efficacy of a proton pump inhibitor (lansoprazole) and a histamine-2 receptor antagonist (famotidine) in preventing recurrent ulcer bleeding in patients with a history of H. pylori-negative idiopathic peptic ulcers.

DETAILED DESCRIPTION:
Peptic ulcer disease used to be caused by a bacterial infection (Helicobacter pylori) in the stomach or the use of certain painkillers (nonsteroidal anti-inflammatory drugs or NSAIDs). However, there has been an increasing trend of peptic ulcer disease with unknown cause (idiopathic ulcer) worldwide since the last decade. Studies in North America found that idiopathic ulcers accounted for 11% and 44% of all peptic ulcers. A meta-analysis of 7 US trials found that 20% of patients with H. pylori-associated ulcers had recurrent ulcers within 6 months, despite successful cure of H. pylori infection and no reported use of NSAIDs. In a pooled analysis of 6 clinical trials with a total of 2900 patients, 27% of duodenal ulcers were not associated with NSAID use or H. pylori infection. The emerging problem of H. pylori-negative idiopathic peptic ulcers is not only limited to western countries. Previously, H. pylori-negative idiopathic peptic ulcers accounted for less than 5% of peptic ulcers in Asia. A recent Korean study reported that the proportion of peptic ulcers not associated with H. pylori infection or NSAID use was over 20%.

ELIGIBILITY:
Inclusion Criteria:

1. A history of H. pylori-negative idiopathic peptic ulcers, defined as

   1. No exposure to aspirin, NSAIDs or drugs of unknown nature including traditional Chinese medicine within the 4 weeks before hospitalization;
   2. Biopsies taken during endoscopy must be negative for both the urease test and histology for H. pylori in the absence of acid suppressive therapy; and
   3. No other causes of ulceration identified.
2. Endoscopically confirmed ulcer healing
3. Age >18 years old
4. Informed consent

Exclusion Criteria:

1. Concomitant steroid or anticoagulant
2. Concomitant use of NSAIDs, aspirin or COX2 inhibitors
3. Previous gastric surgery
4. Requirement of maintenance PPI (e.g. reflux oesophagitis)
5. Advanced comorbidity (defined as ASA 4 or above) or active malignancy
6. Subjects who are pregnant or lactating, or is intending to become pregnant before, during, or within 1 month after participating in this study
7. Subjects who have known hypersensitivity or allergies to any component of lansoprazole or famotidine.
8. Subject who has current or historical evidence of Zollinger-Ellison syndrome or other hypersecretory condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2010-06 (Actual); Primary Completion 2019-05 (Actual); Study Completion 2019-05 (Actual)

PRIMARY OUTCOMES:
Recurrent ulcer bleeding | 24 months
  According to prespecified criteria - hematemesis or melena documented by the admitting physician, or a decrease in the hemoglobin level of at least 2 g/dL, with ulcers or bleeding erosions confirmed on endoscopy.
  A prespecified interim-analysis is performed on the primary endpoint when all patients have been randomised and have completed the 12 months follow-up. The interim-analysis is performed by an independent statistician, blinded for the treatment allocation. The statistician will report to the independent data and safety monitoring committee (DSMC). The DSMC will have unblinded access to all data and will discuss the results of the interim-analysis with the steering committee in a joint meeting. The steering committee decides on the continuation of the trial and will report to the central ethics committee. The Peto approach is used: the trial will be ended using symmetric stopping boundaries at P < 0.001.

SECONDARY OUTCOMES:
Recurrent ulcer detected by endoscopy at 24-month | at the 24th month of follow-up
  Recurrent ulcer detected by endoscopy at 24-month, with or without clinical symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Grace L Wong, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Endoscopy Center, Prince of Wales Hospital, Shatin, Hong Kong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wong GLH, Lau LHS, Ching JYL, Tse YK, Ling RHY, Wong VWS, Chiu PWY, Lau JYW, Chan FKL. Prevention of recurrent idiopathic gastroduodenal ulcer bleeding: a double-blind, randomised trial. Gut. 2020 Apr;69(4):652-657. doi: 10.1136/gutjnl-2019-318715. Epub 2019 Jun 22. PMID 31229990